CLINICAL TRIAL: NCT02192801
Title: Evaluation of Long-term Renal Function in Patients After Surgical Repair of Classical Bladder Exstrophy
Brief Title: Kidney Function in Patients With Bladder Exstrophy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-13-RC-0022-13-CTIL
Record Dates: First submitted 2014-01-30; First posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-01

CONDITIONS: Classic Bladder Exstrophy; Renal Function; GFR; Proteinuria
Keywords: Classic Bladder Exstrophy; Renal function; GFR; Proteinuria
MeSH Terms: conditions — Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with classical bladder exstrophy undergo many surgical interventions with secondary urinary tract infections complicating their course. lately primary definitive surgical correction of this congenital anomaly has been implemented with satisfactory results. Although bladder exstrophy patients are born with normal kidneys, infectious and mechanical surgical complications can potentially damage their kidneys in the long-term. therefore we decided to evaluate renal function in the long-term in these patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients with classic bladder exstrophy treated and followed in Pediatric urology clinic in Dana Children Hospital and Outpatient Clinic

Exclusion Criteria:

* No

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with calssic bladder exstrophy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Renal function | 1 day (last visit )
  Creatinine and GFR estimation , proteinuria, albuminuria will be assessed as measures of renal function as well as renal mass estimation through renal size as by ultrasound and in certain cases through dimercaptosucicnic acid (DMSA)renal scan

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Outpatient Clinic Dana Children Hospital Tel Aviv Sourasky medical center, Tel Aviv, Israel